CLINICAL TRIAL: NCT05352360
Title: Comparison of Pilates Exercises Verses Muscle Energy Techniques Along With Kinesio Taping in Non-Specific Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DPT/Batch-Fall17/517
Record Dates: First submitted 2022-04-14; First posted 2022-04-28 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Pilates Exercises With Kinesio Taping; Muscle Energy Techniques Along With Kinesio Taping

STUDY DESIGN:
Intervention Model Description: This study will help to compare the effects of pilates Exercises with kinesiotaping and on other hand the effects of muscle energy technique with kinesiotaping for improving pain
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pilates Exercises with kinesiotaping (Experimental)
  Interventions: Diagnostic Test: Pilates Exercises
- Muscle energy technique with kinesiotaping (Experimental)
  Interventions: Diagnostic Test: Muscle Energy Technique

INTERVENTIONS:
Diagnostic Test: Pilates Exercises — Exercises with Kinesio Taping
  Arms: Pilates Exercises with kinesiotaping
Diagnostic Test: Muscle Energy Technique — Exercises with Kinesio Taping
  Arms: Muscle energy technique with kinesiotaping

SUMMARY:
To Compare the effects of Pilates Excercises versus muscle energy technique along with kinesiotaping in non specific low back pain.

DETAILED DESCRIPTION:
This study will help to compare the effects of pilates Exercises with kinesiotaping and on other hand the effects of muscle energy technique with kinesiotaping for improving pain, disability and Range of Motion in patient with non specific low back pain. By combining these interventions, time consumption for treatment and disability among community due to low back pain will be reduced. This treatment will be effective for participants for improving function, movement of joints and muscle to manage and treat low back pain. The combination of treatment will be more effective to relief non specific low back pain. The targeted population of 18-40 years old and most of them are having occupational related low back pain or due to bad posture, study will have an impact in improving and managing the low back pain in such population.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of both genders should present with non-specific low back pain and between 18 and 40 years of age.(21)
* Could maintain their standing posture independently for _>30s.
* Patient having enough physical autonomy to participate in the physical activities required by the study.
* The patient having a visual analog scale (VAS) score of equal to or >3 will be included.(16).

Exclusion Criteria:

* A history of spinal surgery, compression fracture, spondylolisthesis, or sciatica, ongoing pregnancy, experiencing hypertension, cardiovascular disease, diabetes mellitus, liver disease, renal disease, rheumatoid arthritis, or other rheumatologically related pathologies (8).
* Those taking corticosteroids 2 weeks before recruitment.
* Hypersensitivity to the tape(6).

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2022-03-31 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Pilates Exercises Verses Muscle Energy Techniques Along with Kinesio Taping | 6 Months
  Comparison of both type of exercises for Non-Specific Low Back Pain

CONTACTS AND LOCATIONS:
Locations (1):
- Chaudhary Muhammad Akram Teaching and research hospital, Jinnah Hospital Lahore and Mayo Hospital Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No